CLINICAL TRIAL: NCT00319488
Title: Childhood Asthma Research and Education (CARE) Network Trial - Acute Intervention Management Strategies (AIMS)
Acronym: AIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Vernon M. Chinchilli, PhD, Pennsylvania State University, College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 386; 5U10HL064313-07 (NIH); 5U10HL064287 (NIH); 5U10HL064307 (NIH); 5U10HL064305 (NIH); 5U10HL064288 (NIH); 5U10HL064295 (NIH)
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2012-04

CONDITIONS: Asthma; Lung Diseases
Keywords: Wheezing; Respiratory Tract Illness
MeSH Terms: conditions — Asthma; Lung Diseases; Respiratory Sounds | interventions — Budesonide; Leukotriene Antagonists; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Active ICS plus placebo LTRA plus albuterol inhalation treatments four times daily
  Interventions: Drug: Inhaled Corticosteroid (Budesonide); Drug: Inhaled Albuterol
- 2 (Active Comparator): Active LTRA plus placebo ICS plus albuterol inhalation treatment four times daily
  Interventions: Drug: Leukotriene Receptor Antagonist (Montelukast Sodium); Drug: Inhaled Albuterol
- 3 (Placebo Comparator): Placebo ICS plus placebo LTRA plus albuterol inhalation treatments four times daily
  Interventions: Drug: Inhaled Albuterol

INTERVENTIONS:
Drug: Inhaled Corticosteroid (Budesonide) — Participants will receive inhaled corticosteroid for 7 days, at the first sign of RTI-associated symptoms.
  Arms: 1
Drug: Leukotriene Receptor Antagonist (Montelukast Sodium) — Participants will receive leukotriene receptor antagonist for 7 days, at the first sign of RTI-associated symptoms.
  Arms: 2
Drug: Inhaled Albuterol — All participants will receive inhaled albuterol treatments four times a day.

SUMMARY:
This study will determine the effectiveness of initiating a high-dose inhaled corticosteroid (ICS) or a leukotriene receptor antagonist (LTRA) in addition to an inhaled beta2-agonist (albuterol) at the onset of respiratory tract illness (RTI)-associated symptoms in increasing episode-free days among young children with recurrent severe wheezing.

DETAILED DESCRIPTION:
Acute Intervention Management Strategies (AIMS) is a randomized, double-blind, double-dummy, placebo-controlled parallel comparison study that will compare the effectiveness of three treatments, when given at the onset of RTI-associated symptoms, in increasing the proportion of symptom-free days over the entire treatment period of the 5- to 9-month study. There will be a 2-week period to qualify and characterize participants, who at that time will have no lower respiratory tract symptoms other than mild cough. A total of 244 participants will be randomized to one of three treatment groups and followed for the remainder of the fall-winter-early spring season. Participants will receive one of the following treatment regimens for 7 days, at the first sign of RTI-associated symptoms: 1) active ICS plus placebo LTRA plus albuterol inhalation treatments four times daily; 2) active LTRA plus placebo ICS plus albuterol inhalation treatment four times daily; or 3) placebo ICS plus placebo LTRA plus albuterol inhalation treatments four times daily.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent episodes (at least two) of wheezing in the context of a RTI, at least one of which must be documented by a health care provider (parental report) over the 12 months prior to study entry, and of which one episode must have occurred within 6 months prior to study entry
* Either two episodes of '1,' OR two episodes of '2,' OR one episode of '1' AND one episode of '2,' defined by the following:

  1. Urgent care visit for acute wheezing (emergency department, urgent care center, or unscheduled primary care physician office visit), which required treatment with a bronchodilator, within 12 months prior to study entry
  2. Episode of wheezing within 12 months prior to study entry, which required treatment with oral corticosteroids not associated with a visit to a health care provider, urgent care center, emergency department, or hospital
* Immunizations are up to date, including varicella (unless the patient has already had clinical varicella)
* Willingness to provide informed consent by patient's parent or guardian

Exclusion Criteria:

* Use of more than six courses of systemic corticosteroids during the 12 months prior to study entry
* More than two hospitalizations for wheezing illnesses within 12 months prior to study entry
* Use of long-term controller medications for asthma (including inhaled corticosteroids, leukotriene modifiers, cromolyn/nedocromil, or theophylline) for 4 or more months (cumulative use) within 1 year prior to study entry
* Any use of long-term controller medications for asthma (including corticosteroids [inhaled or oral], leukotriene modifiers, cromolyn/nedocromil, or theophylline) within the 2 weeks prior to the enrollment visit
* Current treatment with antibiotics for diagnosed sinus disease
* Contraindication of use of systemic corticosteroids
* Prematurity (defined as birth before 36 weeks gestational age)
* Presence of lung disease other than asthma (e.g., cystic fibrosis and BPD)
* Presence of other significant medical illnesses (e.g., cardiac, liver, gastrointestinal, or endocrine disease) that would place the patient at increased risk
* Gastroesophageal reflux under medical therapy
* Immunodeficiency disorders
* History of respiratory failure requiring mechanical ventilation
* History of hypoxic seizure
* Inability to cooperate with nebulization therapy
* Inability to ingest the study drugs
* History of significant adverse reaction to any study medication ingredient
* Current participation, or participation in the month prior to study entry, in another investigational drug study
* Evidence that the family may be unreliable, nonadherent, or likely to move from the clinical center area before study completion
* Persistent symptomatic asthma, as defined as experiencing symptoms (i.e., nocturnal cough, daytime cough, wheezing, difficulty breathing, or symptoms interfering with activities) and/or requiring albuterol use on average 4 or more days per week in the 2-week observation period prior to the randomization visit
* The following scores, based on a 5-point scale with 5 representing very severe symptoms (measured at randomization visit): score equal to or greater than one for albuterol use, wheezing, difficulty breathing, nighttime cough, and asthma symptoms interfering with activities; score greater than 2 for daytime cough on an average of 4 or more days/week during the 2-week observation period
* Failure to complete diary cards at expected levels (at least 80% of days) during the observation period
* Use of long-term controller medications for asthma (e.g., corticosteroids [inhaled or oral], leukotriene modifiers, cromolyn/nedocromil, or theophylline) during the 2-week observation period

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2004-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proportion of episode-free days as determined by diary cards | Measured over 12-month follow-up period

SECONDARY OUTCOMES:
Time to initiation of first course of oral corticosteroids | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Total number of courses of oral corticosteroids | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Duration and severity of lower respiratory tract symptoms | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Number of wheezing episodes | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Time to treatment failure | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Measures of patient and family morbidity | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Number of unscheduled visits for acute wheezing episodes | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization
Linear growth | Measured at Weeks 2, 4, 10, 12, 18, 20, 26, 28, 34, 36, 42, 44, 50, and 52 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Vernon M. Chinchilli, PhD, Principal Investigator — Pennsylvania State University, College of Medicine
Locations (6):
- United States (6):
  - University of Arizona, College of Medicine, Tucson, Arizona
  - UCSD School of Medicine, La Jolla, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Washington University School of Medicine Patient Oriented Research Unit, St Louis, Missouri
  - Dept. of Health Evaluation Sciences, Penn State College of Medicine, Hershey, Pennsylvania
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Result] Bacharier LB, Phillips BR, Zeiger RS, Szefler SJ, Martinez FD, Lemanske RF Jr, Sorkness CA, Bloomberg GR, Morgan WJ, Paul IM, Guilbert T, Krawiec M, Covar R, Larsen G, Mellon M, Moss MH, Chinchilli VM, Taussig LM, Strunk RC; CARE Network. Episodic use of an inhaled corticosteroid or leukotriene receptor antagonist in preschool children with moderate-to-severe intermittent wheezing. J Allergy Clin Immunol. 2008 Dec;122(6):1127-1135.e8. doi: 10.1016/j.jaci.2008.09.029. Epub 2008 Oct 30. PMID 18973936
- [Derived] Fitzpatrick AM, Grunwell JR, Cottrill KA, Mutic AD, Mauger DT. Blood Eosinophils for Prediction of Exacerbation in Preschool Children With Recurrent Wheezing. J Allergy Clin Immunol Pract. 2023 May;11(5):1485-1493.e8. doi: 10.1016/j.jaip.2023.01.037. Epub 2023 Feb 3. PMID 36738927